CLINICAL TRIAL: NCT03562364
Title: Early Advanced Weight Bearing for Peri-articular Knee and Pilon Injuries: An RCT Using the Anti-Gravity Treadmill (AlterG)
Brief Title: Early Advanced Weight Bearing for Peri-articular Knee and Pilon Injuries
Acronym: AlterG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-16-2-0060 AlterG
Record Dates: First submitted 2018-05-15; First posted 2018-06-19 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Distal Femur Fracture; Tibial Plateau Fracture; Distal Tibia Fracture; Pilon Fracture
Keywords: anti-gravity
MeSH Terms: conditions — Femoral Fractures, Distal; Tibial Plateau Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): The standard of care group will remain non-weight bearing for 10-12 weeks following definitive fixation and receive physical therapy in accordance with standard practice at the treating center.
- Early Advanced Weight Bearing (EAWB) (Experimental): The Early Advanced Weight Bearing (EAWB) group will receive early weight-bearing treatment using the antigravity AlterG treadmill. These sessions will begin 14-28 days following definitive fixation and last for a total of 10 weeks
  Interventions: Other: AlterG anti-gravity treadmill

INTERVENTIONS:
Other: AlterG anti-gravity treadmill — The AlterG treadmill is an FDA approved device that allows patients to perform early partial weight bearing exercises in a tightly controlled and safe environment
  Arms: Early Advanced Weight Bearing (EAWB)

SUMMARY:
The overall objective of this study is to compare outcomes following early advanced weight bearing (EAWB) using the AlterG antigravity treadmill versus standard of care physical therapy for adult patients with lower extremity periarticular injuries.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-55
* Closed or Open (Gustilo Type I, II or IIIA) fractures: Distal femur (AO/OTA 33B, 33C), tibial plateau (AO/OTA 41B, 41C), or Distal tibia/pilon (AO/OTA 43B, 43C)
* Definitively treated with a plate
* Ambulatory prior to injury
* Able to participate in rehab starting 28 days after definitive fixation
* Meets AlterG requirements (4'8- 6'4; 85-400lbs)

Exclusion Criteria:

* Medical or psychological disease that would preclude safe functional testing (e.g., severe traumatic brain injury, stroke, heart disease, etc.)
* Prior joint trauma or disease of the operative extremity that resulted in pain, stiffness, or other limitation to mobility
* Injury to the contra-lateral limb, upper extremities or axial skeleton that would influence single limb weight-bearing or use of an assistive device
* Pregnancy
* Unable to speak English
* Severe problems with maintaining follow-up (e.g. patients who are prisoners, homeless at the time of injury, who are intellectually challenged without adequate family support, or have documented psychiatric disorders).
* Unable to provide informed consent.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
The Knee Injury and Osteoarthritis Outcome Score (KOOS) | 6 month following study injury
  The KOOS is a 42 item assessment that evaluates joint function by asking patients to rate their symptoms and concerns in 5 domains: pain, other symptoms, function in daily living (ADL), function in sport and recreation, and foot and ankle quality of life on a scale of 0-4.
Ankle Osteoarthritis Score (AOS) | 6 month following study injury
  The AOS is an assessment that evaluates joint function by asking patients to rate their pain and disability while performing 18 different activities of daily living using a visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Stinner, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (10):
- United States (10):
  - Naval Medical Center San Diego, San Diego, California
  - University of California at San Francisco, San Francisco, California
  - University of Kentucky, Lexington, Kentucky
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Texas Health Science Center - Houston, Houston, Texas
  - San Antonio Military Medical Center (SAMMC), San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Naval Medical Center Portsmouth, Portsmouth, Virginia